CLINICAL TRIAL: NCT02410200
Title: Open-Label, Multicenter, Multiple-Dose Study of the Effect of BG00012 on MRI Lesions and Pharmacokinetics in Pediatric Subjects With Relapsing-Remitting Multiple Sclerosis Aged 10 to 17 Years
Brief Title: Study of the Effect of BG00012 on MRI Lesions and Pharmacokinetics in Pediatric Subjects With RRMS
Acronym: FOCUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109MS202; 2014-005003-24 (EudraCT Number)
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Pediatrics
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BG00012 (Experimental): Oral BG00012 120 mg twice daily (BID) for the first 7 days followed by 240 mg BID for 24 weeks.
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate
  Other Names: BG00012; DMF

SUMMARY:
The primary objective of this study is to evaluate the effect of BG00012 (dimethyl fumarate) on brain magnetic resonance imaging (MRI) lesions in pediatric participants with relapsing-remitting multiple sclerosis (RRMS). The secondary objectives of this study are to characterize the pharmacokinetics of BG00012 in pediatric participants with RRMS and to evaluate the safety and tolerability of BG00012 in pediatric participants with RRMS.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability of parents or legal guardians to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local subject privacy regulations. Subjects will provide assent in addition to the parent or legal guardian, as appropriate, as per local regulations.
* Must have a body weight of ≥30 kg at Screening and Day 1.
* Must have a diagnosis of RRMS according to McDonald criteria for MS (2010) [Polman 2011] and International Pediatric Multiple Sclerosis (MS) Study Group criteria for pediatric MS (2013) [Krupp 2013].

Key Exclusion Criteria:

* Primary progressive, secondary progressive, or progressive relapsing MS (as defined by [Lublin and Reingold 1996]). These conditions require the presence of continuous clinical disease worsening over a period of at least 3 months. Subjects with these conditions may also have superimposed relapses but are distinguished from relapsing-remitting subjects by the lack of clinically stable periods or clinical improvement.
* Disorders mimicking MS, such as other demyelinating disorders (e.g., acute disseminated encephalomyelitis), systemic autoimmune disorders (e.g., Sjögren disease, lupus erythematosus, and neuromyelitis optica), metabolic disorders (e.g., dystrophies), and infectious disorders.
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity to dimethyl fumarate or fumaric acid esters.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (12):
- Research Site, San Bernardino, California, United States
- Research Site, Ghent, Belgium
- Research Site, Sofia, Bulgaria
- Research Site, Hradec Králové, Czechia
- Germany (2):
  - Research Site, München, Bavaria
  - Research Site, Göttingen, Lower Saxony
- Research Site, Dasman, Kuwait City, Kuwait
- Research Site, Riga, Latvia
- Research Site, Beirut, Lebanon
- Poland (2):
  - Research Site, Gdansk
  - Research Site, Poznan
- Research Site, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Alroughani R, Das R, Penner N, Pultz J, Taylor C, Eraly S. Safety and Efficacy of Delayed-Release Dimethyl Fumarate in Pediatric Patients With Relapsing Multiple Sclerosis (FOCUS). Pediatr Neurol. 2018 Jun;83:19-24. doi: 10.1016/j.pediatrneurol.2018.03.007. Epub 2018 Mar 22. PMID 29681490

RESULTS

PARTICIPANT FLOW:
Groups:
- BG00012: BG00012 taken orally at a dose of 120 mg twice daily (BID) for the first 7 days and at a dose of 240 mg BID thereafter for 24 weeks.
Period: Overall Study
Arm/Group | BG00012
Started | 22
Completed | 20
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- BG00012: BG00012 taken orally at a dose of 120 mg BID for the first 7 days and at a dose of 240 mg BID thereafter for 24 weeks.
Arm/Group | BG00012
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (1.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of New or Newly Enlarging T2 Hyperintense Lesions on Brain Magnetic Resonance Imaging (MRI) Scans From the Baseline Period to On-Treatment Assessment Period
Time Frame: Baseline Period (Week -8 to Day 0), On-Treatment Assessment Period (Week 16 to Week 24)
Population: Primary Analysis Population: participants having new or newly enlarging T2 lesions during the Baseline period with a post-baseline assessment.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | BG00012
Number analyzed (Participants) | 15
lesions | -7.9 (16.23)
Statistical Analysis 1: Comparison: BG00012; Test type: Superiority or Other; p = 0.0090, Wilcoxon Signed Rank test

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 8
Population: All participants who received at least 1 dose of BG00012 and had at least 1 pharmacokinetic parameter available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BG00012
Number analyzed (Participants) | 21
ng/mL | 1998.62 (1286.467)

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Day 8
Population: All participants who received at least 1 dose of BG00012 and had at least 1 pharmacokinetic parameter available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BG00012
Number analyzed (Participants) | 21
hours | 4.20 (1.543)

4. Secondary Outcome: Apparent Clearance (CL/F)
Time Frame: Day 8
Population: All participants who received at least 1 dose of BG00012 and had at least 1 pharmacokinetic parameter available.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | BG00012
Number analyzed (Participants) | 17
L/h | 74.45 (30.185)

5. Secondary Outcome: Apparent Volume of Distribution (V/F)
Time Frame: Day 8
Population: All participants who received at least 1 dose of BG00012 and had at least 1 pharmacokinetic parameter available.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | BG00012
Number analyzed (Participants) | 14
L | 98.19 (91.679)

6. Secondary Outcome: Half-Life Lambda z
Time Frame: Day 8
Population: All participants who received at least 1 dose of BG00012 and had at least 1 pharmacokinetic parameter available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BG00012
Number analyzed (Participants) | 14
hours | 0.84 (0.408)

7. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-inf)
Time Frame: Day 8
Population: All participants who received at least 1 dose of BG00012 and had at least 1 pharmacokinetic parameter available.
Measure: Mean (Standard Deviation); unit: h*mcg/mL
Arm/Group | BG00012
Number analyzed (Participants) | 14
h*mcg/mL | 3630.52 (1153.768)

8. Secondary Outcome: Number of Participants Who Experienced Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence that does not necessarily have a causal relationship with treatment. SAE: any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: Up to Week 28
Population: All participants who received at least 1 dose of BG00012.
Measure: Number; unit: participants
Arm/Group | BG00012
Number analyzed (Participants) | 22
participants
  Any event | 20
  Moderate or severe event | 7
  Severe event | 1
  Event related to BG00012 | 16
  Serious event | 5
  Serious event related to BG00012 | 0
  Discontinued treatment due to an event | 2
  Withdrew from study due to an event | 2

ADVERSE EVENTS:
Time Frame: From first dose of study drug through end of treatment period (Week 24 ±7 days) plus 4 weeks follow-up.
Description: Treatment-emergent events are presented.
Arm/Group | BG00012
Serious Adverse Events (participants affected / at risk) | 5/22
Other Adverse Events (participants affected / at risk) | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BG00012 (N=22)
Vertigo (Ear and labyrinth disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BG00012 (N=22)
Vertigo (Ear and labyrinth disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 3
Nasopharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Viral upper respiratory tract infection (Infections and infestations) | 2
Lymphocyte count decreased (Investigations) | 2
Headache (Nervous system disorders) | 4
Multiple sclerosis relapse (Nervous system disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 10
Dysmenorrhoea (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.